CLINICAL TRIAL: NCT05667363
Title: The Effect of a Digital Therapeutics Program on Inhaled Medication Adherence in Patients With Chronic Obstructive Pulmonary Disease：a Prospective, Open-label, Randomized Controlled Clinical Trial
Brief Title: Digital Therapeutics on Inhalation Medication Adherence in COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Ting YANG, MD, PhD, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-HX-43
Record Dates: First submitted 2022-10-24; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Digital Intervention; Inhalation Medication; Adherence
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Intervention (Experimental): Accept metered-dose inhaler medication treatment equipped with digital therapeutics consist of smartphone app and intelligent medication recorder. The intelligent medication recorder can automatically record medication using data and reminds patients through the app. Patients can also record their symptom on the app for doctors to monitor.
  Interventions: Combination Product: Digital Intervention
- Usual use (No Intervention): Accept regular metered-dose inhaler medication treatment.

INTERVENTIONS:
Combination Product: Digital Intervention — Digital therapeutics are consist of a smartphone app and an intelligent medication recorder. The intelligent medication recorder can automatically record medication using data and reminds patients through the app. Patients can also record their symptom on the app for doctors to monitor.
  Arms: Digital Intervention

SUMMARY:
Digital Therapeutics (DTx) is an evidence-based，clinically evaluated software to treat，manage，and prevent a broad spectrum of diseases and disorders according to Digital Therapeutics Alliance，which may improve the adherence of patients with chronic obstructive pulmonary disease (COPD) to use inhaled medication and reduce the risk of acute exacerbation. This study plans to carry out a randomized controlled trial (RCT), using digital therapy to record and manage the behavior data of patients with COPD in the process of using inhaler medication, and analyze the correlation between digital therapy of COPD and patients' drug compliance and treatment effect.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a major disease that causes death and disability worldwide. The World Health Organization (WHO) estimates that COPD has become the third leading cause of death worldwide, accounting for 6% of the global total deaths in 2019. COPD seriously affects the quality of life of patients and causes heavy economic burden to society and families.

Inhaled medication is the key treatment for COPD, and the adherence of inhaled medication is closely related to the effect of disease control. Studies have shown that incorrect and irregular use of metered-dose inhaler are very common in patients.Previous studies have shown that patients using mobile phones to record respiratory symptom diaries, and send blood oxygen saturation, heart rate, body temperature and other data, as well as changes in medication and medical treatment to the portal, and doctors access the data online to identify potential acute exacerbation and take intervention measures, can reduce the risk of acute exacerbation of COPD.

The digital therapeutics of COPD consists of patient mobile phone program, doctor management software and intelligent medication recorder. It develops a digital intervention plan for patients, helping patients intuitively and comprehensively understand the treatment plan and how to act through medication tracking reminder. It also helps doctors to view visualized patient medication, symptoms and other trend data online to understand the real treatment response of patients. This study take digital therapeutics as intervention to explore the correlation between digital therapy and patient medication adherence and treatment effect.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand and willing to sign the written informed consent;
2. Local residents diagnosed COPD by physician;
3. Aged 40 and above;
4. Plan to receive metered-dose inhaler as long-term treatment;
5. Have a smartphone and can apply WeChat applet after training;

Exclusion Criteria:

1. Certain comorbidities (e.g. unstable coronary complications);
2. Undergone thoracic, abdominal or ophthalmic surgery in recent 3 months;
3. Pregnant or lactating women;
4. ABS allergy history.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 582 (Estimated)
Dates: Start 2022-12-20 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of adherent patients. | 24 weeks
  The proportion of patients whose TAI scores 50.

SECONDARY OUTCOMES:
Average times of AECOPD | 4, 12 ,24 weeks
  The average times of self-reported history of AECOPD since the last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ting Yang, MD, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship hospital, Beijing, Beijing Municipality, China